CLINICAL TRIAL: NCT00552838
Title: The Impact of an Antimicrobial Utilization Program on Antimicrobial Use in a Large Public Hospital: A Randomized Controlled Trial
Brief Title: The Impact of an Antimicrobial Utilization Program on Antimicrobial Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 579-2002 Emory IRB
Record Dates: First submitted 2007-10-29; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-09

CONDITIONS: Antimicrobial Prescribing Practices
Keywords: Antimicrobial prescribing; Antimicrobial utilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (No Intervention): Physicians in this arm did not have any intervention with the AUT. Antimicrobial prescriptions were based on hospital guidelines or on the physician's medical knowledge.
  Interventions: Behavioral: Academic Detailing by the Antimicrobial Utilization Team (AUT)

INTERVENTIONS:
Behavioral: Academic Detailing by the Antimicrobial Utilization Team (AUT) — Physicians caring for patients who were prescribed one of three antimicrobials were randomly assigned to academic detailing by the AUT. The AUT would review the antimicrobial prescription and provide consultation to the ordering physician if the prescription is appropriate and provide feedback on a better alternative if inappropriate.

SUMMARY:
Multidisciplinary antimicrobial utilization teams (AUT) have been proposed as an effective mechanism for improving antimicrobial use, but data on their efficacy remain limited. The researchers postulated that a multi-disciplinary AUT would improve antimicrobial use in a teaching hospital when compared to the standard of care (no AUT intervention).

Design: Randomized-controlled intervention trial. Setting: A 953-bed urban teaching hospital.

Patients: Patients admitted to internal medicine ward teams who were prescribed selected antimicrobial agents (piperacillin-tazobactam, levofloxacin, or vancomycin) during the 10month study period.

Intervention: Eight internal medicine ward teams were randomized monthly to academic detailing by the AUT while 8 internal medicine ward teams were randomized indication-based prescription of broad spectrum antimicrobials.

Measurements: Proportion of appropriate empiric, definitive, and end antimicrobial usage (antimicrobial use from the initiation of therapy until definitive therapy is prescribed).

DETAILED DESCRIPTION:
This study was conducted when Bernard C Camins, MD (BCC), one of the investigators, was still employed at Emory University. The principal investigator is no longer at Emory University. This trial is being registered by one of the investigators, BCC, so we can submit the manuscript for publication. BCC is now at Washington University and this study was conducted while he was at Emory University.

ELIGIBILITY:
Inclusion Criteria:

* All patients prescribed vancomycin, piperacillin-tazobactam, or levofloxacin during the time period of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 785 (Actual)
Dates: Start 2002-10; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Appropriateness of Antimicrobial Prescriptions in each group. | 10-month period

SECONDARY OUTCOMES:
Clinical Cure Rate, Mortality Rate between the two groups | 10-month period

CONTACTS AND LOCATIONS:
Overall Officials: Mark D King, MD, MSCR, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Camins BC, King MD, Wells JB, Googe HL, Patel M, Kourbatova EV, Blumberg HM. Impact of an antimicrobial utilization program on antimicrobial use at a large teaching hospital: a randomized controlled trial. Infect Control Hosp Epidemiol. 2009 Oct;30(10):931-8. doi: 10.1086/605924. PMID 19712032